CLINICAL TRIAL: NCT00735124
Title: An Investigation of Post-Operative Pain Scores and Analgesic Requirements After Ambulatory Inguinal Herniorrhaphy With Pre-Operative Gabapentin Therapy
Brief Title: Post-Operative Pain Scores and Analgesic Requirements After Elective Inguinal Herniorrhaphy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Changes to surgical practices led to the loss of eligible patients
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14002
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Pain; Analgesia; Hernia, Inguinal
Keywords: analgesia requirement and post operative pain
MeSH Terms: conditions — Pain; Agnosia; Hernia, Inguinal; Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single pre-op dose of Gabapentine (Active Comparator): Active treatment with the study drug
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo arm for blinding the medication
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Gabapentin — 1200 mg single dose gabapentin
  Other Names: Neurtonin
  Arms: Single pre-op dose of Gabapentine
Other: placebo — Injection of placebo/sham
  Arms: Placebo

SUMMARY:
The study will investigate the effects of single dose pre-operative oral dose of gabapentin (1200) on post -operative pain scores and oral analgesic requirements.

DETAILED DESCRIPTION:
The study will benefit patients in reducing post-operative pain scores as well as reduction in oral analgesic consumption. Gabapentin has been shown to reduce post operative pain pain scores in breast surgery, hysterectomy , spinal surgery, orthopedic and thyroid surgery

ELIGIBILITY:
Inclusion Criteria:

* Subjects having elective surgery with open unilateral Inguinal herniorraphy

Exclusion Criteria:

* Non elective surgery
* Patients currently on gabapentin therapy
* Patient hypersensitive to gabapentin surgery
* History of alcohol or drug abuse
* Patients who are pregnant or who are nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-11-06 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Post operative pain is reduced when single pre-operative oral dose of Gabapentine is given to the patient before the Inguinal Herniorrhaphy | 1yrs
  Post operative pain is reduced when single pre-operative oral dose of

SECONDARY OUTCOMES:
The post operative analgesia requirement is also reduced | 1yrs
  The post operative analgesia requirement is also reduced

CONTACTS AND LOCATIONS:
Overall Officials: Badie Mansour, MD, Principal Investigator — OUHSC
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No